CLINICAL TRIAL: NCT06500585
Title: Effects of Mill's Manipulation Along With Muscle Energy Technique in Lateral Epicondylitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/01788
Record Dates: First submitted 2024-07-08; First posted 2024-07-15 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Lateral Epicondylitis
MeSH Terms: conditions — Tennis Elbow

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mill's Manipulation and Muscle Energy Technique (Experimental): Group A will receive (Mills Manipulation + Muscle Energy Technique + Conventional therapy).
  Interventions: Other: Mill's Manipulation and Muscle Energy Technique
- Mill's Manipulation (Other): Group B will receive (Mills Manipulation + Conventional therapy).
  Interventions: Other: Mill's Manipulation

INTERVENTIONS:
Other: Mill's Manipulation — Mill's Manipulation: The therapist should apply a high-velocity low-amplitude thrust accompanied by a single application . Patients will be treated 3 times a week for 2 consecutive weeks.
  Conventional Therapy:
  Ultrasound therapy: Frequency: 1Mhz Pulse ultrasound: 1:4 Intensity: 1.5 W/cm2 Duration: 5 min.
  Stretching of Wrist Extensors: 15 sec hold, 10 stretches/session/day. Wrist extensors Isometric: resistance 5 to 10 seconds, 15 contractions/ session/day.
  Patients will be treated 3 times a week for 2 consecutive weeks.
  Arms: Mill's Manipulation
Other: Mill's Manipulation and Muscle Energy Technique — Mill's Manipulation:The therapist should apply a high-velocity low-amplitude thrust accompanied by a single application . Patients will be treated 3 times a week for 2 consecutive weeks.
  Muscle Energy Technique: Extensor carpi radialis stretch for 30 sec repeated 5 times during a single treatment session. Patients will be treated 3 times a week for 2 consecutive weeks.
  Conventional Therapy:
  Ultrasound therapy: Frequency: 1Mhz Pulse ultrasound: 1:4 Intensity: 1.5 W/cm2 Duration: 5min.
  Stretching of Wrist Extensors, 15 sec hold, 10 stretches/session/day. Wrist Extensors Isometric, resistance 5 to 10 seconds, 15 contractions/ session/day.
  Patients will be treated 3 times a week for 2 consecutive weeks.
  Arms: Mill's Manipulation and Muscle Energy Technique

SUMMARY:
The effects of Muscle Energy Technique intervention have been investigated in recent studies in Lateral Epicondylitis. Some studies have been conducted about mills manipulation and Muscle Energy Technique but according to the literature review there is no study exist to determine the effects of Mill's Manipulation along with Muscle Energy Technique in Lateral epicondylitis. Because of this reason, further research required to find out the effects of Mill's Manipulation along with Muscle Energy Technique in pain, Range of motion and disability in lateral epicondylitis. So the aim of the study is to determine whether these techniques are effective and should be incorporated frequently in a clinical setting in relation to the conventional therapy. This study will help the clinician for the identification of the better and quick treatment regime which will have no adverse effects and risks and making them more effective, efficient for the patient with lateral epicondylitis.

ELIGIBILITY:
Inclusion Criteria:

* Patient that have been diagnosed with lateral epicondylitis (pain and point tenderness over lateral epicondyle and / or 1-2cm distal to epicondyle).
* Both male and female patients between the age group of 18 to 45 years old.
* Any of the following tests positive: Cozen Test, Mills, Maudsley.

Exclusion Criteria:

* History of rheumatic arthritis
* History of elbow instability
* History of former fracture of the elbow
* History of cervical radiculopathy.
* History of radial tunnel syndrome (Patient with RTS will report pain over lateral forearm approximately 3 to 5 cm distal to the elbow worsens with rotational movements of the forearm).
* History of any neoplasia
* Any congenital or acquired deformity of upper limb.
* History of trauma.
* History of Corticosteroid injection within 6 months.
* Individual having symptoms of vertigo

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2023-10-31 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
NPRS | 2 weeks
  The numeric pain rating scale (NPRS) measure the subjective intensity of pain. NPRS is an eleven point scale from 0 to 10 is the most commonly used version which has good test-retest reliability ( r= .79-.96). The NPRS is a reliable and valid pain assessment scale in LE.
Goniometer | 2 weeks
  Universal goniometer is use to measure wrist ROM in flexion , extension, radial deviation, ulnar deviation, forearm pronation and forearm supination.The intraclass correlation coefficients (ICC) ranged from 0.945 to 0.973 which are classified for the goniometer measurements.
PRFEQ | 2 weeks
  The PRTEE, formerly known as the Patient-Rated Forearm Evaluation Questionnaire (PRFEQ), is a 15-item questionnaire designed to measure forearm pain and disability in patients with lateral epicondylitis (also known as "tennis elbow"). The PRTEE allows patients to rate their levels of tennis elbow pain and disability from 0 to 10, and consists of 2 subscales: 1) PAIN subscale: (0 = no pain, 10 = worst imaginable) Pain - 5 items 2) FUNCTION subscale: (0 = no difficulty, 10 = unable to do) Specific activities - 6 items , Usual activities - 4 items . Test-retest reliability of Korea version PRTEE was good total ICC= .962 (CI=.922-,982). Therefore, it is a useful measure to evaluate the conditions of patients with lateral epicondylitis.

CONTACTS AND LOCATIONS:
Overall Officials: Shamaila Yaqub, Masters, Principal Investigator — Riphah International University
Locations (1):
- Ghosia Medical Centre, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sahoo S, Mohanty RK, Mohapatra J, Equebal A, Das SP. Efficacy of extension wrist hand orthosis on pain, grip strength and electromyographic activities in lateral epicondylitis: A randomized single-blind clinical trial. J Hand Ther. 2023 Oct-Dec;36(4):796-804. doi: 10.1016/j.jht.2023.06.006. Epub 2023 Jul 18. PMID 37474430
- [Background] Kinandana GP, Dewi AANTN, Winaya IMN, Antari NKAJ, Wibawa A, Adhitya IPGS. The Efficacy of Blood Flow Restriction Training for Grip Strength and Disability in Lateral Epicondylitis. Bali Medical Journal. 2023;12(1):410-5.
- [Background] Kucuksen S, Yilmaz H, Salli A, Ugurlu H. Muscle energy technique versus corticosteroid injection for management of chronic lateral epicondylitis: randomized controlled trial with 1-year follow-up. Arch Phys Med Rehabil. 2013 Nov;94(11):2068-74. doi: 10.1016/j.apmr.2013.05.022. Epub 2013 Jun 22. PMID 23796685
- [Background] Bagcaci S, Unuvar BS, Gercek H, Ugurlu I, Sert OA, Yilmaz K. A randomized controlled trial on pain, grip strength, and functionality in lateral elbow pain: Mulligan vs muscle energy techniques. J Back Musculoskelet Rehabil. 2023;36(2):419-427. doi: 10.3233/BMR-220061. PMID 36120766
- [Background] Nambi G, Alghadier M, Verma A, Aldhafian OR, Alshahrani NN, Saleh AK, Omar MA, Hassan TGT, Ibrahim MNA, El Behairy HF. Clinical and radiological effects of Corticosteroid injection combined with deep transverse friction massage and Mill's manipulation in lateral epicondylalgia-A prospective, randomized, single-blinded, sham controlled trial. PLoS One. 2023 Feb 13;18(2):e0281206. doi: 10.1371/journal.pone.0281206. eCollection 2023. PMID 36780557
- [Background] Shukla N, Sharma D, Kumar C, Dixit N. A Comparative Analysis of Effectiveness of Mulligan's Mobilisation Versus Cyriax Approach in the Case of Tennis Elbow. Rivista Italiana di Filosofia Analitica Junior. 2023;14(1):333-41.
- [Background] Cheatham SW, Stull KR, Kolber MJ. Roller massage: is the numeric pain rating scale a reliable measurement and can it direct individuals with no experience to a specific roller density? J Can Chiropr Assoc. 2018 Dec;62(3):161-169. PMID 30662071
- [Background] Khuman PR, Trivedi P, Devi S, Sathyavani D, Nambi G, Shah K. Myofascial release technique in chronic lateral epicondylitis: a randomized controlled study. Int J Health Sci Res. 2013;3(7):45-52.
- [Background] Surangsrirat D, Bualuangngam T, Sri-iesaranusorn P, Chaiyaroj A, Buekban C, Thanawattano C, et al. Comparison of the Wrist Range of Motion Measurement between Inertial Measurement Unit Glove, Smartphone Device and Standard Goniometer. Applied Sciences. 2022;12(7):3418.
- [Background] Armstrong AD, MacDermid JC, Chinchalkar S, Stevens RS, King GJ. Reliability of range-of-motion measurement in the elbow and forearm. J Shoulder Elbow Surg. 1998 Nov-Dec;7(6):573-80. doi: 10.1016/s1058-2746(98)90003-9. PMID 9883416
- [Background] Chapleau J, Canet F, Petit Y, Laflamme GY, Rouleau DM. Validity of goniometric elbow measurements: comparative study with a radiographic method. Clin Orthop Relat Res. 2011 Nov;469(11):3134-40. doi: 10.1007/s11999-011-1986-8. Epub 2011 Jul 21. PMID 21779866
- [Background] Lee D-R, Kim J-S. Reliability and validity of the Korean version of patient-rated tennis elbow evaluation. Journal of Korean Society of Physical Medicine. 2014;9(1):25-33.
- [Background] Kalaskar G, Gurjalwar I, Phansopkar P, Chitale N, Wadhokar OC, Arora SP. Effect of Cyriax physiotherapy and conventional ultrasound on lateral epicondylitis.
- [Background] Saraswati PAS, Thanaya SAP, Nugraha MHS. The Effectiveness Of Dry Needling Versus Muscle Energy Technique Combined With Ultrasound Therapy In Reducing Disability Due To Tennis Elbow. Jurnal Keterapian Fisik. 2022:80-7.
- [Background] Parmar BA, Shukla YU. Effect of eccentric versus concentric exercise on pain, grip strength and function in lateral epicondylitis-a comparative study. Int J Sci Healthcare Res. 2020;5(2):98-109.